CLINICAL TRIAL: NCT07148882
Title: Intranasal Versus Intravenous Fentanyl Effect on Oxidative Stress in Preterm Neonates
Brief Title: Pain Managment in Preterm Neonates
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS683/2023
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-02

CONDITIONS: Preterm Neonates Pain Managment; PreTerm Neonate
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravenous fentanyl (Active Comparator): Intravenous fentanyl group: will receive intravenous fentanyl(1 µg/kg/dose) and typically, one dose is givenMeasure MDA (Malondialdehyde ) level as oxidative stress marker in pain response , venous blood sample 0.5 ml will be collected twice, just before and 30 minutes after the procedure
  Interventions: Drug: fentanyl
- intranasal fentanyl (Active Comparator): Intra nasal fentanyl group: will receive intranasal fentanyl (@fentanyl hamein 50mic/1ml, manufactured by sunny pharmaceutical) using nasal dose of INF is 1.5µg/kg/dose, and typically, one dose is given (Kaushal et al., 2020).
  Measure MDA (Malondialdehyde ) level as oxidative stress marker in pain response , venous blood sample 0.5 ml will be collected twice, just before and 30 minutes after the procedure
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — Intra nasal fentanyl group: will receive intranasal fentanyl using nasal dose of INF is 1.5µg/kg/dose, and typically one dose is given After 5minutes, a second dose could be administrated based on the clinical assessment (maximum two doses per procedure).
  Intravenous fentanyl group: will receive intravenous fentanyl 1 µg/kg/dose and typically, one dose is given After 5minutes, a second dose could be administrated based on the clinical assessment maximum two doses per procedure.
  Measure MDA Malondialdehyde level as oxidative stress marker in pain response , venous blood sample 0.5 ml will be collected twice, just before and 30 minutes after the procedure.
  Monitor adverse events after fentanyl use as apnea cessation of breathing for >20 s, bradycardia heart rate < 100 beats/minute, desaturation oxygen saturation < 80%

SUMMARY:
To compare the effect of Intranasal versus Intravenous Fentanyl on oxidative stress by measuring MDA level just before and after 30 minutes from painful procedure and comparing the results.

DETAILED DESCRIPTION:
1. Intra nasal fentanyl group: will receive intranasal fentanyl using nasal dose of INF is 1.5µg/kg/dose, and typically, one dose is given

   • After 5minutes, a second dose could be administrated based on the clinical assessment (maximum two doses per procedure)
2. Intravenous fentanyl group: will receive intravenous fentanyl(1 µg/kg/dose) and typically, one dose is given •After 5minutes, a second dose could be administrated based on the clinical assessment (maximum two doses per procedure) Measure MDA (Malondialdehyde ) level as oxidative stress marker in pain response , venous blood sample 0.5 ml will be collected twice, just before and 30 minutes after the procedure Monitor adverse events after fentanyl use as apnea (cessation of breathing for >20 s), bradycardia (heart rate < 100 beats/minute), desaturation (oxygen saturation < 80%), and chest wall rigidity associated with laryngospasm (Pacifici, 2015) for 60 min after IN fentanyl administration.

ELIGIBILITY:
Inclusion Criteria:• Preterm neonates during endotracheal intubation

-

Exclusion Criteria:o Contraindication of fentanyl use as hypersensitivity.

* Contraindication of nasal administration of drugs as bilateral occluded nasal passage as choanal atresia and Epistaxis.
* Surgical patients.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
measure MDA level as an oxidative stress marker. | just before fentanyl introduction and half hour after

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams Univercity, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided